CLINICAL TRIAL: NCT04394715
Title: Pragmatic Trial of Messaging to Providers About Treatment of Hyperlipidemia (PROMPT-LIPID)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000027852
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: High Risk Atherosclerotic Cardiovascular Disease
Keywords: electronic alerts; hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Providers will see an electronic alert for eligible patients who are at very high risk for future ASCVD events upon opening of the patient's order entry screen in the medical record.
  Interventions: Other: Electronic Alert
- Control (No Intervention): Providers will not see an electronic alert for any patients and will provide usual care. Silent alerts will be generated that will be sent to study team members.

INTERVENTIONS:
Other: Electronic Alert — Providers will see an automated electronic alert for each eligible hyperlipidemia patient at high risk for future atherosclerotic CVD events. This alert will appear when the provider enters the order entry screen in the patient's medical record during the patient's first eligible outpatient visit. The alert consists of a "pop up" that notifies the physician that the patient is at very high risk for ASCVD events, displays the most recent cholesterol values and the patient's current lipid lowering therapy. It also includes a link to full treatment guidelines for hyperlipidemia, which includes a continuing medical education (CME) option to obtain CME credits.
  Arms: Intervention

SUMMARY:
This study is designed to evaluate the efficacy of automated electronic alerts in the electronic health record to improve rates of best practices in the treatment of patients with hyperlipidemia who present in the setting of outpatient primary care and family medicine practices within the Yale New Haven Health System.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) remains the leading cause of death in most developed countries, including the United States. A key risk factor for CVD is an elevation in low-density lipoprotein cholesterol, or LDL-C. Based on favorable results from large clinical trials, guidelines support the use of high intensity statin therapy for the reduction of LDL-C in very high risk patients and addition of non-statin therapies including ezetimibe and PCSK9 inhibitors if the LDL-C remains above 70 mg/dL. However, implementation of these guidelines is poor and there remains substantial underuse of evidence-based lipid lowering therapies across healthcare systems.

Real-time alerting to important clinical conditions, when fired in an appropriate and timely manner, can have positive impacts on patient outcomes through increased physician awareness and adherence to best practices. To this end, this study has been designed to evaluate whether automated electronic alerts built into the Epic electronic health record can improve the management of hyperlipidemia among patients of outpatient internal medicine and cardiology practices within the Yale New Haven Health System who are at very high risk for future atherosclerotic CVD (ASCVD) events.

One hundred physicians will undergo cluster randomization to either the alert group or the control (usual care) group. Upon opening the order entry screen of an eligible patient with hyperlipidemia, the alert group will receive an informational alert that informs the provider that the patient has hyperlipidemia and is at very high risk for future ASCVD events and provides ACC/AHA-guideline-directed actionable items, including a link to a hyperlipidemia "order set" to include both diagnostic and therapeutic options.

The primary outcome will be the proportion of patients who have intensification of their lipid lowering therapy (increase in statin dose or addition of ezetimibe or addition of a PCSK9 inhibitor) at 90-days. The secondary outcomes will be achieved LDL-C at 6-months and proportion of patients with LDL-C levels less than 70 mg/dL and less than 55 mg/dL. In an optional extension phase, long-term exploratory outcomes looking at the rate of major cardiovascular cardiac events (MACE), defined as hospitalization for myocardial infarction, stroke, unstable angina, or coronary or peripheral artery revascularization will be evaluated at 2 years.

ELIGIBILITY:
Inclusion Criteria for Patient Subjects:

* Adults 18 years of age or greater
* Currently being seen as an outpatient of Internal Medicine or Cardiology within the Yale New Haven Health System
* At very high risk for ASCVD, defined by a history of a major ASCVD event, and most recent lipid profile with LDL-C greater than 70 mg/dL, with or without other high-risk features (diabetes, CKD, age >65 years)

Exclusion Criteria for Patient Subjects:

* Heart transplant recipient
* Left ventricular assist device recipient
* Hospital inpatient status
* Pregnancy
* Have opted out of clinical research in MyChart

Inclusion Criteria for Provider Subjects:

* Practicing at an outpatient cardiology or internal medicine practice with the Yale New Haven Health System
* High frequency of eligible patients seen, based on retrospective review of outpatient records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2596 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nihar Desai, MD MPH, Principal Investigator — Yale University
Locations (4):
- United States (4):
  - Bridgeport Hospotal, Bridgeport, Connecticut
  - Greenwich Hospital, Greenwich, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - St. Raphael's Hospital, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data underlying results for publication will be shared upon publication.
Supporting Information: Study Protocol, SAP
Time Frame: After publication of results; indefinitely

REFERENCES:
- [Derived] Shah NN, Ghazi L, Yamamoto Y, Kumar S, Martin M, Simonov M, Riello Iii RJ, Faridi KF, Ahmad T, Wilson FP, Desai NR. Pragmatic Trial of Messaging to Providers About Treatment of Hyperlipidemia (PROMPT-LIPID): A Randomized Clinical Trial. Circ Cardiovasc Qual Outcomes. 2024 May;17(5):e010335. doi: 10.1161/CIRCOUTCOMES.123.010335. Epub 2024 Apr 18. PMID 38634282
- [Derived] Shah NN, Ghazi L, Yamamoto Y, Martin M, Simonov M, Riello RJ, Faridi KF, Ahmad T, Wilson FP, Desai NR. Rationale and design of a pragmatic trial aimed at improving treatment of hyperlipidemia in outpatients with very high risk atherosclerotic cardiovascular disease: A pragmatic trial of messaging to providers about treatment of hyperlipidemia (PROMPT-LIPID). Am Heart J. 2022 Nov;253:76-85. doi: 10.1016/j.ahj.2022.07.002. Epub 2022 Jul 14. PMID 35841944

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred providers who prescribed the highest volume of PCSK9i in 2020 were retrospectively identified and then consented into the study, followed by randomization into alert group versus usual care group. Patients were automatically enrolled as trial participants if they were seen by a consented provider and met the inclusion criteria as determined by the best practice alert algorithm.
Pre-assignment Details: Four of the 100 providers were excluded from the study before randomization, as recruitment finished before these four providers saw an eligible patient. All 2500 patient subjects were randomized, with zero loss to follow up.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 1179 | 1417
Participants Enrolled | 1130 | 1370
Providers Enrolled | 49 | 47
Completed | 1179 | 1417
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: There were 1130 and 1370 patient subjects enrolled in the alert vs. usual care group, respectively. There were 49 and 47 providers enrolled in the alert vs. usual care group, respectively. The following baseline characteristics are described only for the patient subjects as primary and secondary outcomes were collected only on patient subjects in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 1130 | 1370 | 2500
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 72 [63 to 80] | 71 [62 to 79] | 72 [62 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 531 | 687 | 1218
  Male | 599 | 683 | 1282
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 109 | 132 | 241
  Not Hispanic or Latino | 995 | 1212 | 2207
  Unknown or Not Reported | 26 | 26 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 7
  Asian | 16 | 15 | 31
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 114 | 212 | 326
  White | 890 | 1054 | 1944
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 104 | 86 | 190
Insurance Type [Count of Participants; unit: Participants]
  Medicare | 814 | 974 | 1788
  Medicaid | 294 | 398 | 692
  Commercial | 505 | 582 | 1087
  Other | 254 | 315 | 569
Medical History [Count of Participants; unit: Participants]
  Atrial Arrythmias | 548 | 711 | 1259
  Cerebrovascular Disease | 727 | 1002 | 1729
  Myocardial Infarction | 868 | 1008 | 1876
  Peripheral Artery Disease | 413 | 562 | 975
  Stroke | 555 | 766 | 1321
  Renal Failure | 230 | 299 | 529
  Depression | 246 | 320 | 566
  Diabetes | 353 | 466 | 819
  Hypertension | 988 | 1205 | 2193
  Obesity | 244 | 329 | 573
  Chronic Pulmonary Disorder | 345 | 423 | 768
Baseline Elixhauser Score [Median (Inter-Quartile Range); unit: units on a scale] — This score measures the severity of comorbidities and overall disease burden in hospitalized patients and is used to predict hospital length of stay, hospital charges, and in-hospital mortality. A higher score indicates increased probability of hospital length of stay, resource use, and in-hospital mortality compared to that of a lower score. 21 individual diseases are assigned a weighted score from -7 to 12, and the summation of these scores are used to create the Elixhauser Score, which ranges from -19 (lesser disease burden) to 89 (greater disease burden).
  units on a scale | 5 [3 to 7] | 5 [3 to 8] | 5 [3 to 8]
Cholesterol [Median (Inter-Quartile Range); unit: mg/dL] | 169 [151 to 195] | 172 [152 to 199] | 170 [152 to 197]
HDL [Median (Inter-Quartile Range); unit: mg/dL] | 50 [41 to 61] | 50 [42 to 62] | 50 [41 to 61]
LDL [Median (Inter-Quartile Range); unit: mg/dL] | 91 [78 to 113] | 93 [80 to 117] | 92 [79 to 115]
Triglycerides [Median (Inter-Quartile Range); unit: mg/dL] | 112 [82 to 163] | 112 [82 to 157] | 112 [82 to 159]
AST [Median (Inter-Quartile Range); unit: U/L] | 21 [17 to 28] | 21 [17 to 28] | 21 [17 to 28]
ALT [Median (Inter-Quartile Range); unit: U/L] | 20 [15 to 29] | 21 [15 to 29] | 21 [15 to 29]
Creatinine [Median (Inter-Quartile Range); unit: mg/dL] | 1 [.84 to 1.23] | .96 [.8 to 1.2] | 1 [.8 to 1.2]
Baseline Blood Pressure [Median (Inter-Quartile Range); unit: mmHg]
  Systolic BP | 130 [119 to 140] | 129 [120 to 140] | 129 [120 to 140]
  Diastolic BP | 74 [68 to 80] | 74 [68 to 80] | 74 [68 to 80]
Baseline Heart Rate [Median (Inter-Quartile Range); unit: beats/minute] | 72 [64 to 82] | 72 [64 to 80] | 72 [64 to 81]
Baseline Number of Lipid Lowering Therapy (LLT) Medications [Median (Inter-Quartile Range); unit: Number of medications] | 1 [.25 to 1] | 1 [1 to 1] | 1 [1 to 1]
Number of subjects on Lipid Lowering Therapy Medications [Count of Participants; unit: Participants]
  Any statin | 803 | 982 | 1785
  Low intensity statin | 37 | 52 | 89
  Moderate intensity statin | 278 | 330 | 608
  High intensity statin | 488 | 600 | 1088
  Ezetimibe | 85 | 134 | 219
  PCSK9i | 28 | 38 | 66
Patients per Provider Type [Count of Participants; unit: Participants]
  Cardiology Physician | 730 | 785 | 1515
  Cardiology Advanced Practice Provider | 68 | 118 | 186
  Internal Medicine Physician | 280 | 280 | 560
  Internal Medicine Advanced Practice Provider | 52 | 187 | 239

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Intensification of Lipid Lowering Therapy
Description: Intensification of lipid lowering therapy is defined as an increase in statin dose, an addition of ezetimibe, or addition of PCSK9. Any one of the three will be sufficient to meet this endpoint. Proportion of patients who meet this endpoint will be compared between study arms.
Time Frame: 90 days from first alert for any given patient
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1130 | 1370
Participants | 159 | 142

2. Secondary Outcome: Achieved LDL-C at 6 Months
Description: LDL-C at 6 months as measured by medical record review
Time Frame: 6 months from first alert for any given patient
Population: This outcome was only observed in 824 patient subjects in which data for LDL-C at 6 months was available. 368 patient subjects in the intervention arm and 456 patient subjects in the control arm received 6 month LDL-C measurements that were placed in the medical record, thus this is the population analyzed for this outcome.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Intervention | Control
Number analyzed (Participants) | 368 | 456
mg/dL | 83 [66.5 to 102] | 83 [68 to 107]

3. Secondary Outcome: Proportion of Patients With an LDL-C of Less Than 70 mg/dL
Description: Number of patients with LDL-C levels less than 70 mg/dL based on medical record review. Number of patients who meet this endpoint will be compared between study arms.
Time Frame: 6 months from first alert for any given patient
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 368 | 456
Participants | 115 | 133

4. Secondary Outcome: Proportion of Patients With an LDL-C of Less Than 55 mg/dL
Description: Number of patients with LDL-C levels less than 55 mg/dL based on medical record review. Number of patients who meet this endpoint will be compared between study arms.
Time Frame: 6 months from first alert for any given patient
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 368 | 456
Participants | 45 | 53

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events are reported to the IRB via written report within 5 calendar days of the Principal Investigator becoming aware of the event.
  Adverse events reporting is only described for patient subjects as the exposure of interest would be expected to affect this study population. Adverse events were not monitored or assessed for provider subjects.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 18/1130 | 29/1370
Serious Adverse Events (participants affected / at risk) | 0/1130 | 0/1370
Other Adverse Events (participants affected / at risk) | 0/1130 | 0/1370

LIMITATIONS AND CAVEATS:
All study sites were in a single academic health system, and the alert was developed within this site's EHR, reducing generalizability. The study relied on accurately documented ASCVD ICD-10 codes. Contamination between providers at shared sites was possible, biasing the outcome toward the null. Finally, many providers chose to defer the alert, suggesting responsibility of LLT intensification belonged to primary care providers or cardiologists.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT04394715/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/15/NCT04394715/ICF_001.pdf